CLINICAL TRIAL: NCT04483895
Title: Comparison Between the Oro-Helical Length Technique and the 7-8-9 Rule in Determination of the Ideal Endotracheal Tube Insertion Depth in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Mohamed Shinkar, Assistant professor of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Maha Abdel-Raouf master thesis
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The OHL method (Active Comparator): the ETT insertion depth was estimated according to the OHL method.
  Interventions: Procedure: Endotracheal tube insertion
- The 7-8-9 method (Active Comparator): the ETT insertion depth was estimated according to the 7-8-9 method.
  Interventions: Procedure: Endotracheal tube insertion

INTERVENTIONS:
Procedure: Endotracheal tube insertion — ETT was inserted and the depth was estimated by either OHL method or 7-8-9 method

SUMMARY:
This study was conducted on neonates needing intubation; Group A,: the ETT insertion depth was estimated according to the OHL method. Group B,: the ETT insertion depth was estimated according to the 7-8-9 method.

ELIGIBILITY:
Inclusion Criteria:

* • Full term and preterm neonates who were admitted to NICU and needing endotracheal intubation for invasive mechanical ventilation or administration of surfactant.

  * Delivery room intubations were not included as infants are not routinely weighed prior to resuscitation at our hospital. However, infants intubated in the delivery room who were subsequently intubated in the NICU were eligible for inclusion in our study.

Exclusion Criteria:

- 1. Major upper or lower airway anomalies. 2. Infants with craniofacial, vertebral anomalies. 3. Significant congenital anomalies including cardiac, abdominal or respiratory.

4. Neonates those whose parents declined consent were excluded from the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-12-21 (Estimated); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
the proportion of ETTs in abnormal position for each of both insertion depth prediction methods. | 28 days

SECONDARY OUTCOMES:
the occurrence of pulmonary air leaks during the first 24 hours after intubation, accidental extubation and duration of ventilation. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- medicine -Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided